CLINICAL TRIAL: NCT06168552
Title: Exploratory Clinical Study of Fluorescent Navigation Technology Based on Anti-EGFR Antibody-IR800CW Novel Imaging Agent in Radical Resection of Pancreatic Cancer
Brief Title: Fluorescent Navigation Technology in Radical Resection of Pancreatic Cancer
Acronym: CISPD-6
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, The chairman of the First Affiliated Hospital of Zhejiang University School of Medicine, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CISPD-6
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Resectable Pancreatic Adenocarcinoma
Keywords: resectable pancreatic cancer; Fluorescence navigation technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): The patient underwent Da Vinci robot or fluorescent laparoscopic-assisted radical resection of pancreatic cancer. The day before the operation, anti-EGFR antibody-IR800CW imaging agent was injected into the vein, and the fluorescence test was performed to evaluate the imaging of the primary lesions of the pancreas and the intra-abdominal lymph nodes. And to evaluate for the presence of imaging lesions in the liver, peritoneum, pelvic cavity, etc.
  Interventions: Diagnostic Test: Injection of fluorescent developer (anti-EGFR-IR800CW)

INTERVENTIONS:
Diagnostic Test: Injection of fluorescent developer (anti-EGFR-IR800CW) — The patient underwent Da Vinci robot or fluorescent laparoscopy-assisted radical resection of pancreatic cancer, and anti-EGFR antibody-IR800CW imaging agent was injected in the day before surgery, and fluorescence detection was performed

SUMMARY:
This study intends to design the prospective, exploratory, single center clinical study, using targeted EGFR fluorescence imaging agent (anti-EGFR-IR800CW) and fluorescent navigation technology, in its lymph node tracing, intraoperative tumor localization, accurate determination of resection margin, and explore its clinical significance in radical surgical resection of pancreatic cancer.

DETAILED DESCRIPTION:
The overall prognosis of pancreatic cancer is poor. For resectable patients, adjuvant chemotherapy is performed after surgery, which has become the standard and standard treatment recommended by various guidelines. Preoperative neoadjuvant therapy is proved to improve the R0 resection rate and reduce the lymph node metastasis rate, thus prolonging the postoperative recurrence-free survival time and increasing the survival benefit of patients. But despite adequate preoperative and postoperative treatment, the patient benefit remains limited. In pancreatic cancer surgery, improving the R0 resection rate, increasing the positive lymph node resection rate, and accurately identifying small metastases to accurately stage, can improve the prognosis of patients to a certain extent. Therefore, this study intends to design the prospective, exploratory, single center clinical study, using targeted EGFR fluorescence imaging agent (anti-EGFR-IR800CW) and fluorescent navigation technology, in its lymph node tracing, intraoperative tumor localization, accurate determination of resection margin, and explore its clinical significance in radical surgical resection of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined the study and signed the informed consent form; Age is greater than or equal to 18 years old (time for signing the informed consent form);
2. Minimally invasive radical surgical resection can be performed after discussion and evaluation of hepatobiliary and pancreatic surgery;
3. The patient and his family members volunteered to receive radical surgical resection of pancreatic cancer; Patients must have reliable contraception during the study and within 6 months after the study period;
4. negative serum pregnancy / urine pregnancy test within 7 days before study enrollment and must be non-lactating subjects;
5. male subjects should agree to have contraception during the study and within 6 months after the end of the study period;

Exclusion Criteria:

1. Combined diseases and medical history:

1. Severe organ failure, such as respiratory failure, uncontrolled thyroid dysfunction including hyperthyroidism and hypothyroidism, or uncorrection of K +, Na +, Ca 2 + electrolyte disorders;
2. Within 5 years, the subject had previous or both other malignant tumors (except for cured skin basal cell carcinoma and cervical carcinoma in situ); with other malignant tumors, but the following two conditions were enroll: other malignant tumors treated with single surgery with R0 resection and no recurrence for 5 years; cured cervical carcinoma in situ, skin basal cell carcinoma, nasopharyngeal carcinoma and superficial bladder tumor [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];

2. There are surgical contraindications;

3. Study Treatment-Related to:

1. Previous history of severe allergy to macromolecular drugs, or allergy to known ingredients of EGFR injection;
2. Chronic treatment with systemic hormones or other immunosuppressive agents (dose> 10mg / day prednisone or other efficacy hormone) 28 days prior to the start of the study and continued hormone or immunosuppressive agents within 2 weeks after the first test administration, immunomodulators included: therapeutic vaccines, cytokine therapy, or subjects against CTLA 4,4-1BB, OX-40 (except for regular use, temporary);
3. Active autoimmune diseases requiring systemic treatment (e. g., corticosteroids or immunosuppressants) occurred within 2 years prior to the initiation of study treatment. Alternative therapies (e. g. thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency, etc.) are not considered as systemic therapy;

4. According to the discretion of the investigator, subjects with serious hazards to subject safety or concomitant diseases completing the study, or no other reasons for the enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy and sensitivity of the imaging agent | 1 month after enrolled
  Accuracy and sensitivity of anti-EGFR antibody-IR800CW imaging technology of primary pancreatic lesions and metastatic lymph nodes in radical resection of pancreatic cancer

IPD SHARING:
Plan to Share IPD: No